CLINICAL TRIAL: NCT02642367
Title: Comparison of With or Without Use of Stylet for Endotracheal Intubation With McGrath Videolaryngoscope
Brief Title: Stylet Use for McGrath Videolaryngoscope
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jong Yeop Kim, Associate profefssor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AJIRB-MED-DE4-15-345
Record Dates: First submitted 2015-12-22; First posted 2015-12-30 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Orotracheal Intubation
MeSH Terms: interventions — Rocuronium

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- no use of stylet (Experimental): Endotracheal intubation was performed 2 min after rocuronium injection without use of stylet with McGrath videolaryngoscope after endotracheal tube was rolled up circularly for 3 min
  Interventions: Device: McGrath videolaryngoscope; Drug: rocuronium
- use of stylet (Active Comparator): Endotracheal intubation was performed 2 min after rocuronium injection using a styletted endotracheal tube with McGrath videolaryngoscope
  Interventions: Device: McGrath videolaryngoscope with Intubating stylet (Mallinckrodt); Drug: rocuronium

INTERVENTIONS:
Device: McGrath videolaryngoscope — without use of stylet
  Arms: no use of stylet
Device: McGrath videolaryngoscope with Intubating stylet (Mallinckrodt) — use of stylet
  Arms: use of stylet
Drug: rocuronium — tracehal intubation was performed 2 min after rocuronium injection with McGrath videolaryngoscope
  Other Names: rocumeron

SUMMARY:
The routine use of a styletted endotracheal tube during videolaryngoscopy is advocated by some manufacturers, but styletted endotracheal tube can elicit rare but potentially serious complications. We compared the intubation time and success rate whether or not use of stylet for endotracheal intubation with McGrath videolaryngoscope.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status I or II undergoing orotracheal intubation for elective surgery

Exclusion Criteria:

* cervical spine injury
* rapid sequence induction
* body mass index> 35 kg/m2
* airway pathology

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2016-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
intubation time | 2 min after rocuronium injection
  time the blade passed the lips until endtidal CO2 was detected

CONTACTS AND LOCATIONS:
Overall Officials: Jong Yeop Kim, Study Director — Ajou University School of Medicine
Locations (2):
- South Korea (2):
  - Ajou University Hospital, Suwon, Gyeongki-do
  - Ajou University Hospital, Suwon